CLINICAL TRIAL: NCT00642512
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Efficacy Study of Oral Dronabinol Alone and in Combination With Ondansetron Versus Ondansetron Alone in Subjects With Delayed Chemotherapy-Induced Nausea and Vomiting
Brief Title: Dronabinol Versus Standard Ondansetron Antiemetic Therapy in Preventing Delayed-Onset Chemotherapy-Induced Nausea and Vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Vickie Baranowski, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S175.3.102
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-03

CONDITIONS: Chemotherapy Induced Nausea and Vomiting
Keywords: CINV; chemotherapy; nausea; vomiting; retching
MeSH Terms: conditions — Vomiting; Nausea | interventions — Dronabinol; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: dronabinol
- 2 (Active Comparator)
  Interventions: Drug: ondansetron
- 3 (Other)
  Interventions: Drug: dronabinol/ondansetron
- 4 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dronabinol — 10 - 20 mg
  Arms: 1
Drug: ondansetron — 8 - 16 mg
  Arms: 2
Drug: dronabinol/ondansetron — 10 - 20 mg/8 - 16 mg
  Arms: 3
Drug: placebo — placebo
  Arms: 4

SUMMARY:
The primary purpose of the study is to determine the efficacy of oral dronabinol versus standard ondansetron antiemetic therapy in preventing delayed-onset chemotherapy-induced nausea and vomiting (CINV) or retching by measuring the incidence of total response of nausea and vomiting and/or retching following administration of moderate-to-high emetogenic chemotherapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

* Histological evidence of non-CNS malignancy (primary or metastatic disease) and lymphomas which are not involving the bone marrow.
* Undergoing single or multiple days of chemotherapy as long as Day 1 chemotherapy includes:

  1. a moderate-to-high emetogenic regimen, or
  2. oxaliplatin at doses employed for treatment of colon cancer, or
  3. the combination of AC [AdriamycinÒ (60 mg/m2) with cyclophosphamide (600 mg/m2)] as to be used for the chemotherapeutic drug regimen involving taxanes in the treatment of breast cancer.

Exclusion Criteria:

* Chemotherapy agents falling into the low (Level 1), moderate-to-low (Level 2), moderate (Level 3) unless used in combination with a Level 4 chemotherapy agent on Day 1 of the study.
* Chemotherapy agents falling into the high (Level 5) classification during study.
* Any combination of chemotherapy agents that does not fall into the moderate-to-high (Level 4) classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2003-07; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Total response of nausea and vomiting/retching was defined as no vomiting and/or retching, an intensity of nausea of < 5 mm on the visual analog scale (VAS) and no use of rescue medication. | 5 days

SECONDARY OUTCOMES:
Complete responder rate (no vomiting/retching, intensity of nausea of ≤ 30 mm on the VAS and no use of rescue medication) | 5 days
Presence or absence of nausea | 5 days
Episodes of vomiting and/or retching | 5 days
Duration of nausea and vomiting and/or retching | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (43):
- United States (43):
  - Site 970, Tucson, Arizona
  - Site 950, Anaheim, California
  - Site 925, Fountain Valley, California
  - Site 913, Greenbrae, California
  - Site 909, Los Angeles, California
  - Site 908, Pomona, California
  - Site 943, Rancho Mirage, California
  - Site 932, Boynton Beach, Florida
  - Site 924, Hollywood, Florida
  - Site 940, Lakeland, Florida
  - Site 921, New Port Richey, Florida
  - Site 929, New Port Richey, Florida
  - Site 933, Ormond Beach, Florida
  - Site 922, Marietta, Georgia
  - Site 928, Harvey, Illinois
  - Site 914, Orland Park, Illinois
  - Site 926, Skokie, Illinois
  - Site 946, Springfield, Illinois
  - Site 956, Terre Haute, Indiana
  - Site 905, Southfield, Michigan
  - Site 916, Fergus Falls, Minnesota
  - Site 937, Greenwood, Mississippi
  - Site 958, St Louis, Missouri
  - Site 904, Missoula, Montana
  - Site 919, Little Silver, New Jersey
  - Site 920, Voorhees Township, New Jersey
  - Site 948, Brooklyn, New York
  - Site 953, Brooklyn, New York
  - Site 910, The Bronx, New York
  - Site 949, Valhalla, New York
  - Site 947, Wilmington, North Carolina
  - Site 902, Bismarck, North Dakota
  - Site 942, Fargo, North Dakota
  - Site 944, Columbus, Ohio
  - Site 934, Oklahoma City, Oklahoma
  - Site 931, Philadelphia, Pennsylvania
  - Site 906, Pittsburgh, Pennsylvania
  - Site 918, Charleston, South Carolina
  - Site 923, North Charleston, South Carolina
  - Site 917, Chattanooga, Tennessee
  - Site 939, Chattanooga, Tennessee
  - Site 915, Texarkana, Texas
  - Site 951, Arlington, Virginia